CLINICAL TRIAL: NCT01845701
Title: Phase III Study to Study the Clinical Response to ACT Fixed Dose Combination in 42 Days in Uncomplicated Malaria in Cameroon
Brief Title: Artemisinin-Based Antimalarial Combinations and Clinical Response in Cameroon
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Yaounde 1 (Other)
Collaborators: World Health Organization (Other); Gates Malaria Partnership (Other)
Responsible Party: Principal Investigator, Wilfred F. Mbacham, ScD, PI, University of Yaounde 1
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A60041
Record Dates: First submitted 2013-04-28; First posted 2013-05-03 (Estimated); Last update posted 2018-09-26 (Actual); Status verified 2018-09

CONDITIONS: Malaria
Keywords: malaria, cure rate, efficacy, safety
MeSH Terms: conditions — Malaria | interventions — amodiaquine, artesunate drug combination; Artemether, Lumefantrine Drug Combination

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Artesunate-Amodiaquine (Experimental): As a fixed-dose combination of artesunate-amodiaquine developed by Sanofi-Aventis (France). It has the advantage of being a 3-day regimen usable by all age groups and potentially low cost. tablets are administered per every day at dose of 25mg/67.5mg for those between 4,5kg and 9kg for 48H
  Interventions: Drug: Artesunate-Amodiaquine
- Dihydroartemisinine_Piperaquine (Experimental): As a fixed-dose combination of dihydroartemisinin-piperaquine which is produced by Fouley (China). It is a potentially low cost 2-day regimen that has been used in children between 5-10kg as half a tablet of 40mg/320mg every day for 48H
  Interventions: Drug: Dihydroartemisinine-Piperaquine
- Artemeter-Lumefantrine (Active Comparator): This is the active comparator as a fixed-dose combination of artemether and lumefantrine which is produced by Novartis (Switzerland). The drug will be used as the comparator because it is the only fixed-dose combination with artemether currently available. Administered in children as tablets containing Artemether-Lumefantrine at (20mg/120mg) for body weights of 5-10kg every 12H within 48H.
  Interventions: Drug: Artemether-lumefantrine combination

INTERVENTIONS:
Drug: Artesunate-Amodiaquine — Pharmacology: Amodiaquine is effective against the erythrocytic stages of all four species of P. falciparum. Amodiaquine accumulates in the parasite's lysosomes and prevents breakdown of haemoglobin on which the parasite depends for its survival.
  Artesunate is a water-soluble hemisuccinate derivative of artemisinin. Artesunate and its active metabolite dihydroartemisinin are potent blood schizonticides, active against the ring stage of the parasite.
  The fixed-dose combination dihydroartemisinin-piperaquine has a cost advantage over other ACTs that brings it within reach of many, making it a potential best candidate for deployment in Africa and other poor countries. The drug is currently produced in China (Duo-cotecxin®).
  Other Names: CoArsucam
  Arms: Artesunate-Amodiaquine
Drug: Dihydroartemisinine-Piperaquine — It is a bisquinoline antimalarial drug (1,3-bis[1-(7-chloro-4 quinolyl)-4- piperazinyl]-propane) that was first synthesised in the 1960s, and used extensively in China and Indochina as prophylaxis and treatment during the next 20 years. A number of Chinese research groups documented that it was at least as effective as, and better tolerated than, chloroquine against falciparum and vivax malaria. With the development of piperaquine-resistant strains of P. falciparum and the emergence of the artemisinin derivatives, its use declined during the 1980s. However, during the next decade, piperaquine was rediscovered by Chinese scientists as one of a number of compounds suitable for combination with an artemisinin derivative.
  Other Names: Duo-Cotecxin
  Arms: Dihydroartemisinine_Piperaquine
Drug: Artemether-lumefantrine combination — CoArtem® is an oral, fixed combination of artemether- a derivative of artemisinin and lumefantrine- a novel molecule developed by the Academy of Military Medical Sciences (AMMS) in Beijing. It is the only co-formulated ACT approved by WHO and is currently available through WHO at a negotiated public sector price. Both compounds are effective as single agents. However, recrudescence is common with artemether and lumefantrine has a slow onset of action. A fixed combination tablet (20 mg artemether/120 mg lumefantrine) has therefore been developed. Fixed combination therapy improves compliance and has the advantage of carrying a lower risk of selecting drug resistant strains. No resistance to either component has been observed to date.
  Other Names: CoArtem
  Arms: Artemeter-Lumefantrine

SUMMARY:
To assess the efficacy of artesunate-amodiaquine, dihydroartemisinin-piperaquine, in comparison with artemether-lumefantrine during 42 days follow up period in 720 children with acute uncomplicated P. falciparum malaria, in two different endemic ecological areas - Savanna and equatorial forest regions of Cameroon.

We have set as specific objectives:

* To assess the efficacy of artesunate-amodiaquine, dihydroartemisinin-piperaquine, in comparison with artemether-lumefantrine during 14 and 28 days follow up period in children with acute uncomplicated P. falciparum malaria in two different endemic areas.
* To evaluate the safety of artesunate-amodiaquine, dihydroartemisinin-piperaquine, in comparison with artemether-lumefantrine during 42 days follow up period in children with acute uncomplicated P. falciparum malaria.
* To determine parasite clearance time (PCT) and fever clearance time (FCT) following the administration of the three trial regimens.
* To investigate the treatment response based on WHO criteria (WHO, 2003) in patients in all groups after trial.
* To investigate the Single Nucleotide Polymorphisms (SNPs) and microsatellite markers of genes associated with drug resistance

DETAILED DESCRIPTION:
Methodology Children of either gender, between 6 months (> 5kg) and 10 years of age, with acute uncomplicated P. falciparum infection, who fulfil all of the inclusion and have none of exclusion criteria will be enrolled in the study. They will be randomised to receive the three trial arms, i.e, Study Arm-A: artesunate-amodiaquine, Study Arm-B: dihydroartemisinin-piperaquine and Study Arm-C: artemether-lumefantrine at the ratio of 2:2:1 and will be hospitalised over a 3-day period to facilitate the supervised administration of the study drugs and full clinical and laboratory assessment and observation of early adverse effects. On discharge, participants will be required to report to the study clinic on days 7, 14, 21,28, 35 and 42 or at any other time when clinical sign(s)/symptom(s) of malaria is suspected. The number of participants is about 720 children

Inclusion Criteria

* Children of either gender, aged between 6 months (> 5kg) and 10 years.
* Suffering from acute uncomplicated P. falciparum malaria confirmed by microscopy using Giemsa-stained thick film with an asexual parasite density of 1,000 to 100,000 parasites/μl.
* Presenting with fever (axillary temperature ≥ 37.5oC) or having a history of fever in the preceding 24 hours.
* Able to ingest tablets orally (either suspended in water or uncrushed with food).
* Willing to participate in the study with written assent from parent/guardian. Parental authorization will be obtained for children less than 8 years old and documented assent of parents/guardians for children 8-10 years.
* Willing and able to attend the clinic on stipulated regular follow-up visits.

Exclusion Criteria

• Any of the following "danger signs of severe malaria": Not able to drink or breast feed Persistent vomiting (>2 episodes within previous 24 hours) Convulsions (>1 episode within previous 24 hours) Lethargic/unconscious

* Signs/symptoms indicating severe/complicated malaria according to WHO criteria (WHO definition).
* Concomitant illnesses, underlying chronic hepatic or renal disease, abnormal cardiac rhythm, hypoglycaemia, jaundice, respiratory distress,
* Serious gastrointestinal disease, severe malnutrition (W/H < 70%) or severe anaemia (haemoglobin < 5 g/dl).
* Known hypersensitivity to the study drugs.

ELIGIBILITY:
Inclusion Criteria:

* Children of either gender, aged between 6 months (> 5kg) and 10 years.
* Suffering from acute uncomplicated P. falciparum malaria confirmed by microscopy using Giemsa-stained thick film with an asexual parasite density of 1,000 to 100,000 parasites/μl.
* Presenting with fever (axillary temperature ≥ 37.5oC) or having a history of fever in the preceding 24 hours.
* Able to ingest tablets orally (either suspended in water or uncrushed with food).
* Willing to participate in the study with written assent from parent/guardian. Parental authorization will be obtained for children less than 8 years old and documented assent of parents/guardians for children 8-10 years.
* Willing and able to attend the clinic on stipulated regular follow-up visits.

Exclusion Criteria:

•Any of the following "danger signs of severe malaria": Not able to drink or breast feed Persistent vomiting (>2 episodes within previous 24 hours) Convulsions (>1 episode within previous 24 hours) Lethargic/unconscious

* Signs/symptoms indicating severe/complicated malaria according to WHO criteria (WHO definition).
* Concomitant illnesses, underlying chronic hepatic or renal disease, abnormal cardiac rhythm, hypoglycaemia, jaundice, respiratory distress,
* Serious gastrointestinal disease, severe malnutrition (W/H < 70%) or severe anaemia (haemoglobin < 5 g/dl).
* Known hypersensitivity to the study drugs.

Ages: 6 Months to 120 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 720 (Actual)
Dates: Start 2010-03; Primary Completion 2014-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Clinical Efficacy | 42 days
  Patient's trial outcome will be classified according to the WHO guidelines (WHO 2003) with application as follows: Early Treatment Failure (ETF); Late Clinical Failure (LCF); Late Parasitological Failure (LPF); Adequate Clinical and Parasitological Response (ACPR) - Absence of parasitaemia on day 42 irrespective of temperature without previously meeting any of the criteria of early treatment failure or late clinical failure or late parasitological failure

SECONDARY OUTCOMES:
Safety by measure of changes in Physiologic, Blood, Liver and Kidney functions to define AE & SAEs | 42 days
  Prevalence of adverse events (AEs) and serious adverse events (SAEs): proportion of patients who experience AEs or SAEs during the follow up period of 42 days.
  Changes in vital Physiologic parameters (blood pressure, pulse rate): proportion of patients who have significant changes in vital signs comparing to baseline during the follow up period of 42 days.
  Prevalence of abnormal laboratory tests: proportion of patients who have abnormal values of laboratory tests (ALAT, ASAT, Bilirubin, Creatinine, Glucose, Urea etc), during the follow up period of 42 days.

CONTACTS AND LOCATIONS:
Overall Officials: Wilfred F Mbacham, ScD, Principal Investigator — University of Yaounde 1
Locations (2):
- Cameroon (2):
  - L'Hopital de District Ngong, Garoua,, Garoua, North Region
  - Baptist Hospital, Mutengene, South-West Region

REFERENCES:
- [Derived] Nji AM, Ali IM, Moyeh MN, Ngongang EO, Ekollo AM, Chedjou JP, Ndikum VN, Evehe MS, Froeschl G, Heumann C, Mansmann U, Ogundahunsi O, Mbacham WF. Randomized non-inferiority and safety trial of dihydroartemisin-piperaquine and artesunate-amodiaquine versus artemether-lumefantrine in the treatment of uncomplicated Plasmodium falciparum malaria in Cameroonian children. Malar J. 2015 Jan 28;14:27. doi: 10.1186/s12936-014-0521-2. PMID 25626448